CLINICAL TRIAL: NCT03562793
Title: Communication and Activation in Pain to Enhance Relationships and Treat Pain With Equity (COOPERATE)
Brief Title: Communication and Activation in Pain to Enhance Relationships and Treat Pain With Equity
Acronym: COOPERATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 17-032; 1712397218 (Other: Indiana University)
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-03

CONDITIONS: Pain
Keywords: pain; healthcare disparities; communication
MeSH Terms: conditions — Pain; Communication

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with behavioral intervention.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to treatment assignment when administering baseline outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COOPERATE Intervention Arm (Experimental): Intervention patients will focus on 1) goal clarification/prioritization; 2) communication skills. There are 6 total sessions delivered individually over 12 weeks: 4 sessions teaching skills (30 min each) and 2 booster sessions delivered once/month for the next 2 months. Intervention will be delivered by telephone.
  Interventions: Behavioral: Communication and Activation in Pain to Enhance Relationships and Treat Pain with Equity (COOPERATE)
- Attention Control Arm (No Intervention): Veterans randomized to the control group will receive phone calls on the same schedule as intervention Veterans. During these phone calls, study staff will ask Veterans a series of questions about their pain, self-management activities, and any changes they have experienced since the last call. These phone calls are designed to control for attention only, and Veterans will not be offered specific information or advice about their pain or its management (with the exception of suggesting a doctor visit if warranted).

INTERVENTIONS:
Behavioral: Communication and Activation in Pain to Enhance Relationships and Treat Pain with Equity (COOPERATE) — . COOPERATE seeks to improve patient activation in minority Veterans with chronic pain by focusing on two major skill sets: 1) goal clarification and prioritization, and 2) communication skills (Table 1). By understanding, clarifying, and prioritizing goals, and having the skills to communicate their goals, priorities, and preferences to providers, Veterans will gain knowledge, confidence, and skills to be actively involved in managing their chronic pain. The intervention consists of 6 total sessions delivered individually over 12 weeks: 4 sessions focused on teaching skills related to goal clarification/prioritization and communication (30-minutes each), delivered weekly for the first 4 weeks, plus 2 booster sessions (20-25 minutes each) delivered once per month for the next 2 months.
  Other Names: COOPERATE
  Arms: COOPERATE Intervention Arm

SUMMARY:
Chronic pain affects approximately 100 million Americans and 40-70% of Veterans, and amounts to over $600 billion/year in direct medical costs and lost worker productivity. Racial disparities in pain care are well-documented, within and outside VA. Minorities are more likely to be undertreated for pain, are subjected to more urine drug tests, and are referred for substance abuse evaluation more frequently than Whites. Minority patients also exhibit lower levels of engagement and active involvement in their healthcare, which leads to poorer communication with providers and poorer outcomes. COOPERATE is a randomized controlled trial testing an intervention to improve minority Veterans' active participation in their pain care by focusing on 2 essential skill sets: 1) goal-setting and prioritization, and 2) communication skills.

DETAILED DESCRIPTION:
Background: Chronic pain affects 40-70% of Veterans and amounts to over $600 billion/year in direct medical costs and lost worker productivity. Racial disparities in pain treatment have been extensively documented. Minority patients, including Veterans, are more likely to be undertreated for pain. Minority Veterans have pain documented less frequently, undergo more urine drug tests, and are more likely to be referred for substance abuse evaluation than White Veterans. Compounding these pain care disparities, minority Veterans exhibit lower levels of patient activation than Whites. Patient activation-having knowledge, confidence, and skills to manage health-is associated with better health experiences, self-management, and outcomes. Low activation is frequently manifested in poorer communication among minority patients. Minority patients are less likely to share their concerns with providers, ask questions, and prepare for their clinic visits. This poor communication is associated with lower quality care, poorer patient-provider relationships, and treatment non-adherence. The poorer communication experienced by minorities is exacerbated by the documented difficulties in patient-provider communication about chronic pain and its treatment-particularly where opioids are concerned.

Objectives: COOPERATE (Communication and Activation in Pain to Enhance Relationships and Treat Pain with Equity) is a pragmatic randomized controlled trial of an intervention to improve patient activation and communication with providers for minority Veterans with chronic pain. COOPERATE focuses on 2 essential skill sets necessary to facilitate effective patient activation: 1) goal-setting and prioritization, and 2) communication skills. COOPERATE is delivered over the telephone in 6 sessions (4 weekly sessions followed by 2 booster session) over a period of 12 weeks. The primary study outcome is patient activation.

Methods: COOPERATE is a Hybrid Type 1 study, designed to test effectiveness while also examining implementation facilitators and barriers. COOPERATE will enroll 250 minority Veterans with chronic musculoskeletal pain from primary care clinics. Veterans will be randomized either to the COOPERATE intervention or to an attention control arm. For Aim 1 the investigators will test the effects of COOPERATE at 3 (primary end point), 6, and 9 months (sustained effects) on patient activation (primary outcome), communication self-efficacy, pain intensity and interference, and psychological functioning. In Aim 2, the pre-implementation aim, the investigators will use qualitative methods to understand facilitators and barriers to implementing COOPERATE. Guided by the RE-AIM framework, the investigators will interview a purposefully selected subsample of intervention Veterans, and clinicians from primary care and the chronic pain clinic, to better prepare for COOPERATE's implementation. Aim 3 is an exploratory aim to determine the effects of COOPERATE on important relational indicators of high-quality care: working alliance (with providers), and perceived discrimination in healthcare.

Innovation: COOPERATE focuses on two important, yet frequently neglected, areas for improvement in minority health: patient activation and communication. This is especially important in chronic pain care, since numerous treatment options with a wide range of risks and benefits exist, and since minorities are offered fewer of these pain treatment options. Helping minority Veterans to become more active in their care is critical for improving chronic pain care. This is especially important in light of VA efforts such as the Opioid Safety Initiative, designed to improve safety for Veterans, but which also require engaged, active patients as Veterans must explore alternative pain treatments with their providers-treatments that are feasible for Veterans' individual lifestyles and consistent with their symptom priorities and treatment goals.

ELIGIBILITY:
Inclusion Criteria:

* Black or African American Veteran
* Have musculoskeletal pain in the low back, cervical spine, or extremities (hip, knee, shoulder) for 3 months

Exclusion Criteria:

Patients will be excluded if electronic medical records indicate:

* a psychotic disorder diagnosis
* current substance use disorder
* severe medical conditions precluding participation (e.g., NY Heart Association Class III or IV heart failure), or if the eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Sassi Matthias, PhD MS BA, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Matthias MS, Hirsh AT, Ofner S, Daggy J. Exploring the Relationships Among Social Support, Patient Activation, and Pain-Related Outcomes. Pain Med. 2022 Apr 8;23(4):676-685. doi: 10.1093/pm/pnab306. PMID 34718764
- [Result] Matthias MS, Adams J, Burgess DJ, Daggy J, Eliacin J, Flores P, Hirsh AT, Myers LJ, Perkins AJ, Menen T, Procento P, Rand KL, Salyers MP, Shanahan ML, Bair MJ. Communication and Activation in Pain to Enhance Relationships and Treat Pain with Equity (COOPERATE): Rationale, study design, methods, and sample characteristics. Contemp Clin Trials. 2022 Jul;118:106790. doi: 10.1016/j.cct.2022.106790. Epub 2022 May 12. PMID 35568376
- [Result] Matthias MS, Adams J, Burgess D, Daggy J, Eliacin J, Flores P, Hirsh AT, Myers LJ, Perkins AJ, Menen T, Philip Procento, Rand KL, Salyers MP, Shanahan ML, Bair MJ. Corrigendum to: Communication and Activation in Pain to Enhance Relationships and Treat Pain with Equity (COOPERATE): Rationale, study design, methods, and sample characteristics (Contemporary Clinical Trials, volume 118, article number 106790). Contemp Clin Trials. 2022 Sep;120:106883. doi: 10.1016/j.cct.2022.106883. Epub 2022 Aug 20. No abstract available. PMID 35999166
- [Result] Matthias MS, Adams J, Burgess DJ, Daggy J, Gowan TM, Perkins AJ, Eliacin J. Effects of the COVID-19 Pandemic on Black Veterans' Mental Health: A Qualitative Investigation. J Health Care Poor Underserved. 2022;33(3):1275-1290. doi: 10.1353/hpu.2022.0112. PMID 36245163
- [Result] Matthias MS, Burgess DJ, Eliacin J. Healthcare Access and Delivery During the COVID-19 Pandemic for Black Veterans with Chronic Pain: a Qualitative Study. J Gen Intern Med. 2023 Mar;38(4):1024-1029. doi: 10.1007/s11606-022-07884-9. Epub 2022 Nov 14. PMID 36376625
- [Derived] Matthias MS, Daggy JK, Perkins AJ, Adams J, Bair MJ, Burgess DJ, Eliacin J, Flores P, Myers LJ, Menen T, Procento P, Rand KL, Salyers MP, Shanahan ML, Hirsh AT. Communication and activation in pain to enhance relationships and treat pain with equity (COOPERATE): a randomized clinical trial. Pain. 2024 Feb 1;165(2):365-375. doi: 10.1097/j.pain.0000000000003021. Epub 2023 Sep 21. PMID 37733487

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Started | 124 | 126
3 Months | 103 | 120
6 Months | 100 | 113
Completed | 99 | 104
Not Completed | 25 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm | Total
Number analyzed (Participants) | 124 | 126 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Overall study population is 250. There were 126 randomized to the control group and 124 randomized to the intervention group.
  years | 61.3 (10.1) | 60.6 (9.9) | 61.0 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Overall study population is 250. There were 126 randomized to the control group and 124 randomized to the intervention group.
  Participants
    Female | 19 | 24 | 43
    Male | 105 | 102 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall study population is 250. There were 126 randomized to the control group and 124 randomized to the intervention group.
  Participants
    Hispanic or Latino | 1 | 2 | 3
    Not Hispanic or Latino | 123 | 124 | 247
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Overall study population is 250. There were 126 randomized to the control group and 124 randomized to the intervention group.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 124 | 126 | 250
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 124 | 126 | 250

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation
Description: Patient Activation Measure (PAM). Construct: self-management self-efficacy (i.e., patient activation). 13-item patient activation measure assesses patient knowledge, skill, and confidence for self-management. Range 0 (lowest activation) - 100 (highest activation). Higher values are better outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 103 | 120
units on a scale | 60.39 (13.55) | 57.58 (13.51)

2. Primary Outcome: Patient Activation
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 100 | 113
units on a scale | 62.82 (15.96) | 58.18 (13.97)

3. Primary Outcome: Patient Activation
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 124 | 126
units on a scale | 55.69 (13.92) | 57.45 (13.07)

4. Primary Outcome: Patient Activation
Description: as for outcome 1
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 99 | 104
units on a scale | 61.56 (14.13) | 58.56 (12.64)

5. Secondary Outcome: Communication Self-Efficacy (Perceived Efficacy in Patient-Physician Interactions--PEPPI)
Description: Perceived Efficacy in Patient-Physician Interactions (PEPPI-5). Construct: patients' self-efficacy in obtaining medical info and getting most important concerns discussed with their doctors. Range 0 (lowest) - 50 (highest). Higher values are better outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 103 | 120
units on a scale | 38.27 (9.63) | 36.65 (10.81)

6. Secondary Outcome: Pain Intensity and Interference (Brief Pain Inventory)
Description: Brief Pain Inventory (BPI). Construct: Pain Intensity and Interference. 11-item measure that assesses pain intensity and interference with activity. The Brief Pain Inventory (BPI) assesses two key domains-intensity and interference-recommended for pain studies and has been validated in primary care. The BPI is the average of pain intensity and pain interference scores. The pain intensity score is an average of 4 ratings of 0 (no pain) to 10 (pain as bad as you can imagine) for current, least, worst, and average pain in the past week. The pain interference score averages seven ratings, 0 (does not interfere) to 10 (interferes completely), of interference with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Lower scores are better outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 103 | 120
units on a scale | 5.02 (2.45) | 5.31 (2.28)

7. Secondary Outcome: Depression (PHQ8)
Description: Patient Health Questionnaire (PHQ)-8. Construct: Depression. Validated 8-item measure assessing depression severity. Range 0 - 24. Lower scores are better outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 103 | 120
units on a scale | 8.50 (5.79) | 9.08 (5.86)

8. Secondary Outcome: Anxiety
Description: GAD 7. Construct: Anxiety. Validated 7-item measure to assess anxiety. Range 0 - 21. Lower scores are better outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 103 | 120
units on a scale | 6.70 (5.77) | 7.21 (6.03)

9. Secondary Outcome: Pain Coping
Description: Coping Strategies Questionnaire. Construct: Pain coping. A 14-item measure of pain coping strategies. Range 0-84. Lower scores are better outcomes.
Time Frame: Change from baseline to 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 103 | 120
units on a scale | 14.42 (5.94) | 13.91 (5.60)

10. Secondary Outcome: Communication Self-Efficacy (Perceived Efficacy in Patient-Physician Interactions--PEPPI)
Description: as for outcome 5
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 124 | 126
units on a scale | 34.64 (11.30) | 35.73 (10.56)

11. Secondary Outcome: Communication Self-Efficacy (Perceived Efficacy in Patient-Physician Interactions--PEPPI)
Description: as for outcome 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 100 | 113
units on a scale | 39.41 (9.69) | 37.90 (9.06)

12. Secondary Outcome: Communication Self-Efficacy (Perceived Efficacy in Patient-Physician Interactions--PEPPI)
Description: as for outcome 5
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 99 | 104
units on a scale | 39.46 (9.67) | 37.98 (9.11)

13. Secondary Outcome: Pain Intensity and Interference (Brief Pain Inventory)
Description: as for outcome 6
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 124 | 126
units on a scale | 5.67 (2.15) | 5.35 (2.11)

14. Secondary Outcome: Pain Intensity and Interference (Brief Pain Inventory)
Description: as for outcome 6
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 100 | 113
units on a scale | 5.19 (2.41) | 5.10 (2.37)

15. Secondary Outcome: Pain Intensity and Interference (Brief Pain Inventory)
Description: as for outcome 6
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 99 | 104
units on a scale | 5.46 (2.38) | 5.02 (2.35)

16. Secondary Outcome: Depression (PHQ8)
Description: as for outcome 7
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 124 | 126
units on a scale | 8.82 (5.64) | 8.14 (5.68)

17. Secondary Outcome: Depression (PHQ8)
Description: as for outcome 7
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 100 | 113
units on a scale | 8.33 (5.90) | 8.69 (6.02)

18. Secondary Outcome: Depression (PHQ8)
Description: as for outcome 7
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 99 | 104
units on a scale | 8.87 (6.16) | 8.87 (5.76)

19. Secondary Outcome: Anxiety
Description: GAD 7. Construct: Anxiety. Validated 7-item measure to assess anxiety. Range 0 - 21. Lower scores are better outcomes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 124 | 126
units on a scale | 7.37 (5.79) | 6.66 (5.61)

20. Secondary Outcome: Anxiety
Description: GAD 7. Construct: Anxiety. Validated 7-item measure to assess anxiety. Range 0 - 21. Lower scores are better outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 100 | 113
units on a scale | 7.07 (6.01) | 7.04 (6.18)

21. Secondary Outcome: Anxiety
Description: GAD 7. Construct: Anxiety. Validated 7-item measure to assess anxiety. Range 0 - 21. Lower scores are better outcomes.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
Number analyzed (Participants) | 99 | 104
units on a scale | 7.11 (6.32) | 7.14 (5.66)

ADVERSE EVENTS:
Time Frame: 9 months
Description: Adverse events were documented by research staff.
Groups:
- COOPERATE Intervention Arm: No adverse events.
  Intervention patients will focus on 1) goal clarification/prioritization; 2) communication skills. There are 6 total sessions delivered individually over 12 weeks: 4 sessions teaching skills (30 min each) and 2 booster sessions delivered once/month for the next 2 months. Intervention will be delivered by telephone.
  Communication and Activation in Pain to Enhance Relationships and Treat Pain with Equity (COOPERATE): . COOPERATE seeks to improve patient activation in minority Veterans with chronic pain by focusing on two major skill sets: 1) goal clarification and prioritization, and 2) communication skills (Table 1). By understanding, clarifying, and prioritizing goals, and having the skills to communicate their goals, priorities, and preferences to providers, Veterans will gain knowledge, confidence, and skills to be actively involved in managing their chronic pain. The intervention consists of 6 total sessions delivered individually over 12 weeks: 4 sessions focused on teaching skills related to goal clarification/prioritization and communication (30-minutes each), delivered weekly for the first 4 weeks, plus 2 booster sessions (20-25 minutes each) delivered once per month for the next 2 months.
- Attention Control Arm: No adverse events.
  Veterans randomized to the control group will receive phone calls on the same schedule as intervention Veterans. During these phone calls, study staff will ask Veterans a series of questions about their pain, self-management activities, and any changes they have experienced since the last call. These phone calls are designed to control for attention only, and Veterans will not be offered specific information or advice about their pain or its management (with the exception of suggesting a doctor visit if warranted).
Arm/Group | COOPERATE Intervention Arm | Attention Control Arm
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/126
Other Adverse Events (participants affected / at risk) | 0/124 | 0/126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03562793/Prot_SAP_000.pdf